CLINICAL TRIAL: NCT06710444
Title: Ultrasound-guided Erector Spinae Plane Block Versus Retrolaminar Block for Postoperative Analgesia in Patients Undergoing Percutaneous Nephrolithotomy
Brief Title: Erector Spinae Plane Block Versus Retrolaminar Block for Analgesia in Percutaneous Nephrolithotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Shehab, MD, Lecturer in Anaesthesia and Surgical ICU department, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0306627
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Analgesia; Pain Management; PCNL; Regional Anesthesia Block
Keywords: Postoperative; Analgesia; Pain; Erector Spinae; Retrolaminar; Block; PCNL
MeSH Terms: conditions — Agnosia; Pain; Bites and Stings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Active Comparator): This group will receive ultrasound-guided erector spinae plane block
  Interventions: Procedure: ultrasound-guided erector spinae plane block
- Group II (Experimental): This group will receive ultrasound-guided Retrolaminar plane block
  Interventions: Procedure: ultrasound-guided retrolaminar plane block

INTERVENTIONS:
Procedure: ultrasound-guided erector spinae plane block — ESPB
  Arms: Group I
Procedure: ultrasound-guided retrolaminar plane block — RLB
  Arms: Group II

SUMMARY:
The study will investigate the effects of ultrasound-guided ESPB and RLB on intraoperative and postoperative analgesia in patients undergoing PCNL to identify a safe and effective regional block method for postoperative analgesia

DETAILED DESCRIPTION:
All the patients will be blinded to the intervention received in this study. All patients will receive standard general anesthesia technique with endotracheal intubation and muscle paralysis. Postoperatively, all patients will receive analgesia in the form of non-steroidal anti-inflammatory drugs and paracetamol. In case the VAS scores exceeded 4 in any group, the patients will receive rescue analgesia with 25 mg IV meperidine. In both groups, the ESPB and RLB will be performed after induction of general anesthesia using portable ultrasound device.

ELIGIBILITY:
Inclusion Criteria:

- Patients scheduled for PCNL

Exclusion Criteria:

* daily consumption of analgesics
* allergy to local anesthetics
* liver dysfunction
* infection or previous surgery in the vertebral region.
* patient refusal
* pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
measurement of visual analogue score | after the surgery average 48 hours postoperative
  measurement of visual analogue score during rest and movement. The Score range from 0-10. 0 means no pain and 10 indicates the worst pain ever

SECONDARY OUTCOMES:
postoperative additional analgesic requirement | after the surgery average 48 hours postoperative
  Total cumulative analgesic requirement dose
assessing the patient satisfaction by a the short assessment of patient satisfaction score (SAPS) | after the surgery average 48 hours postoperative
  from 0 to 28, where 0 is so dissatisfied and 28 means very satisfied
Time to ambulate | after the surgery average 12 hours postoperative
  Time from discharge from the operating theatre to start to ambulate
presence of postoperative nausea and vomiting | after the surgery average 48 hours postoperative
  Number of postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S. Shehab, MD, Principal Investigator — Alexandria University
Locations (1):
- Ahmed S.Shehab, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: Yes
there is a plan to make individual participant data (IPD) collected in this study, including data dictionaries, available to other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After study ends upon request
Access Criteria: Accessible through the web site

REFERENCES:
- [Background] Sotome S, Sawada A, Wada A, Shima H, Kutomi G, Yamakage M. Erector spinae plane block versus retrolaminar block for postoperative analgesia after breast surgery: a randomized controlled trial. J Anesth. 2021 Feb;35(1):27-34. doi: 10.1007/s00540-020-02855-y. Epub 2020 Sep 11. PMID 32915300